CLINICAL TRIAL: NCT06318351
Title: Observing the Influence of Transcutaneous Acupoint Electrical Stimulation on Postoperative Delirium After Thoracoscopic Lung Resection Surgery - a Multicenter Cohort Study
Brief Title: Transcutaneous Acupoint Electrical Stimulation and Postoperative Delirium Delirium
Status: Recruiting | Type: Observational
Sponsor: Qin Zhang (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Qin Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202402015
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Delirium, Postoperative
Keywords: Delirium; Thoracoscopic lung resection surgery
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transcutaneous Electrical Acupoint Stimulation: The effect of Transcutaneous Electrical Acupoint Stimulation on postoperative vision was observed according to anesthesiologist's habit of using or not using it.
  Interventions: Procedure: transcutaneous acupoint electrical stimulation

INTERVENTIONS:
Procedure: transcutaneous acupoint electrical stimulation — This is a safe and non-invasive procedure, similar to an electrode sheet, which applies a weak current to a specific site to achieve the purpose of acupoint stimulation.

SUMMARY:
Investigating postoperative delirium in patients undergoing thoracoscopic lung resection surgery who have received or not received relevant transcutaneous acupoint electrical stimulation treatment preoperatively, observing postoperative recovery quality indicators, evaluating the necessity of treatment, and clarifying the potential mechanisms by which transcutaneous acupoint electrical stimulation may improve postoperative delirium.

DETAILED DESCRIPTION:
Research design type: multicenter, prospective, cohort observational trial. The leading unit is Tongji Hospital affiliated with Tongji Medical College of Huazhong University of Science and Technology, and the participating unit is Guangdong Provincial Hospital of Chinese Medicine (a large comprehensive traditional Chinese medicine hospital directly under the National Administration of Traditional Chinese Medicine), skilled in using traditional Chinese medicine treatment methods to improve postoperative recovery quality. Participating in a multicenter clinical study on transcutaneous acupoint electrical stimulation to improve postoperative delirium after thoracoscopic surgery will help collectively explore the perioperative application and mechanism of action of traditional Chinese medicine techniques for acupoint stimulation.

Firstly, patients meeting the inclusion criteria from the Department of Thoracic Surgery of Tongji Hospital affiliated with Tongji Medical College of Huazhong University of Science and Technology and Guangdong Provincial Hospital of Chinese Medicine will be recruited. Upon admission, the Mini-Mental State Examination (MMSE) will be used as a routine clinical assessment to screen all patients for cognitive status to reduce the impact of cognitive impairments on subsequent observations. Subsequently, based on whether patients receive transcutaneous acupoint electrical stimulation treatment by an anesthesiologist, patients will be divided into two groups (yes or no for receiving the treatment). Their recovery period, delirium assessment within 7 days postoperatively, as well as assessments of sleep, pain, etc., will be observed. Preoperative and postoperative peripheral blood samples will be collected for testing related indicators. Information on demographic characteristics, discharge diagnosis, laboratory indicators at admission and discharge, postoperative complications, length of hospital stay, disease awareness, etc., will be collected from the medical records system for statistical analysis to explore the correlation between transcutaneous acupoint electrical stimulation and postoperative delirium in patients undergoing thoracoscopic lung resection.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the study;
2. Age ≥ 18 years;
3. Patients scheduled for thoracoscopic lung resection surgery;
4. ASA grade I-III.

Exclusion Criteria:

1. History of severe central nervous system diseases, psychiatric disorders, cognitive impairment, intellectual disability, or Mini-Mental State Examination (MMSE) score ≤23;
2. History of opioid addiction, long-term use of analgesic drugs, or psychotropic drugs;
3. Severe cardiovascular and cerebrovascular diseases;
4. Severe liver and kidney dysfunction: Child-Pugh grade B, C patients, patients requiring regular dialysis, etc.;
5. Pregnant or postpartum women;
6. Patients with language communication barriers;
7. Deemed unsuitable for participation by the researchers.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing thoracoscopic pneumonectomy
Sampling Method: Probability Sample
Enrollment: 476 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Delirium | 7days
  Mini-Mental State Examination, MMSE

SECONDARY OUTCOMES:
Recovery | 7days
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Qin Zhang, phd, Principal Investigator — Tongji Medical College, Huazhong University of Science and Technology
Locations (2):
- China (2):
  - Guangdong Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei